CLINICAL TRIAL: NCT01449045
Title: Cluster Randomized Trial of Malaria Seasonal IPTc Combined With Community Case Management in Saraya District, SE Senegal
Brief Title: Trial of Malaria Seasonal IPTc Combined With Community Case Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cheikh Anta Diop University, Senegal (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Jean Louis Ndiaye, Assistant Professor, Cheikh Anta Diop University, Senegal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SEN11.16; TA.2010.40200.032 (Other Grant/Funding Number: EDCTP)
Record Dates: First submitted 2011-09-11; First posted 2011-10-07 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Malaria
Keywords: IPTc; Community Case Management; Home Management for malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community Case Management (Placebo Comparator): Provision of access to prompt diagnosis and treatment for malaria by community volunteers in the village (PECADOM)
  Interventions: Drug: Community Case Management with artemether-lumefantrine (AL)
- Community Case Management plus IPTc (Experimental): Monthly Intermittent Preventive Treatment with sulfadoxine pyrimethamine plus amodiaquine, in addition to community case management
  Interventions: Drug: IPTc+CCM

INTERVENTIONS:
Drug: IPTc+CCM — Monthly administration of sulfadoxine-pyrimethamine plus amodiaquine, combined with community case management
  Arms: Community Case Management plus IPTc
Drug: Community Case Management with artemether-lumefantrine (AL) — Malaria diagnosis with Rapid Diagnostic Test and treatment with AL if the test is positive
  Arms: Community Case Management

SUMMARY:
Malaria is a major public health problem. 250 million cases annually leads to approximately 1 million deaths. Over 80 per cent of these deaths occur among African children under age five. The main interventions covered treatment with Artemisinin Combination Therapies (ACT), long lasting bednets distribution and Rapid Diagnosis Tests (RDT) to improve malaria diagnosis. This has led in Senegal to a substantial decrease in the incidence of malaria, in 2009. However the recent overall decline hides the fact that malaria incidence remains very high in the south of Senegal. That's why Home-based management (HMM) for malaria is being introduced in selected areas. Intermittent Preventive Treatment (IPT) by monthly administration of a therapeutic dose of antimalarials can achieve a very high degree of protection from attacks of clinical malaria in children. The purpose of this project is to evaluate the effectiveness of combining IPTc with HMM in southern Senegal

The study objectives are to :

* Assess the tolerance of IPTc using SP+AQ when it is administered for a longer period in areas with a longer transmission season,
* Assess the added benefit that IPT with the association of Sulfadoxine-Pyrimethamine + Amodiaquine can offer in populations where a rapid and early care with home management of malaria is already established.
* Determine the cost benefit ratio of the addition of IPTc with HMM. A cluster randomized controlled trial has been designed to evaluate the effectiveness of adding seasonal IPTc with sulfadoxine-pyrimethamine plus amodiaquine (SP+AQ) for 5 months per year, in villages where home-based management of malaria is implemented. All villages in Saraya district, excluding 7 villages with a health post, will be eligible to participate. Saraya villages will be combined to form 24 clusters which will be randomized to receive HMM from a community volunteer, or IPTc plus HMM. Trained volunteer Community Medicine Distributors (CMD) will provide HMM. The primary endpoint will be the incidence of clinical malaria with fever or history of fever and parasitaemia with density of at least 3000/ul. Secondary outcomes will include the safety, the tolerability, the coverage and acceptability of the intervention. Both the recurrent and capital costs to the health service of training staff and delivering the interventions will be estimated. Both direct and indirect costs to users of the services (children and their families) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age between 3 to 120 months
* consent participation given by parents or guardians
* willing to remain in the study area in the next 6 months

Exclusion Criteria:

* Known allergy to the study investigational drug
* Any underlying chronic or severe condition.
* Participant under Treatment with sulfamides

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4554 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of children under 10 years of age with clinical malaria | up to 24 weeks
  children under 10 years age presenting symptoms of malaria with fever (or history of fever in the previous 48 hours) with a positive Rapid Diagnostic Test or positive blood slides

SECONDARY OUTCOMES:
Number of children under 10 years of age presenting clinical Malaria with high parasite density | up to 24 weeks
  Malaria with parasite density at 3000 parasites/uL or more in the presence of fever or history of fever in the previous 48hours in children under 10 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Oumar Gaye, PhD, Study Director — Cheikh Anta Diop University, Senegal; Paul Milligan, PhD, Study Chair — London School of Hygiene and Tropical Medicine; Badara Cisse, PhD, Study Chair — Cheikh Anta Diop University, Senegal
Locations (1):
- University Cheikh Anta Diop, Dakar, Senegal

REFERENCES:
- [Derived] Ndiaye JLA, Ndiaye Y, Ba MS, Faye B, Ndiaye M, Seck A, Tine R, Thior PM, Atwal S, Beshir K, Sutherland C, Gaye O, Milligan P. Seasonal malaria chemoprevention combined with community case management of malaria in children under 10 years of age, over 5 months, in south-east Senegal: A cluster-randomised trial. PLoS Med. 2019 Mar 13;16(3):e1002762. doi: 10.1371/journal.pmed.1002762. eCollection 2019 Mar. PMID 30865632